CLINICAL TRIAL: NCT01836549
Title: A Molecular Biology and Phase II Study of Imetelstat (GRN163L) in Children With Recurrent High-Grade Glioma, Ependymoma and Diffuse Intrinsic Pontine Glioma
Brief Title: Imetelstat Sodium in Treating Younger Patients With Recurrent or Refractory Brain Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to several intracranial hemorrhages and recommendation by the PBTC DSMB.
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-036; NCI-2013-00482 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01CA081457 (NIH)
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-06

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Ependymoma; Astrocytoma, Grade II; Ependymoma; Giant Cell Glioblastoma; Glioblastoma; Gliosarcoma; Oligodendroglioma; Brainstem Tumors
MeSH Terms: conditions — Astrocytoma; Ependymoma; Glioblastoma; Gliosarcoma; Oligodendroglioma; Brain Stem Neoplasms | interventions — imetelstat; GRN163L peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (imetelstat sodium) (Experimental): Molecular Biology Phase: Patients will receive one infusion of imetelstat prior to surgery. Surgery will take place 12-24 hours after the infusion of imetelstat. Patients will continue to receive therapy on the same schedule as the Phase II patients starting 14-21 days after surgery.
  Phase II: Patients receive imetelstat sodium IV over 2 hours on days 1 and 8. Treatment repeats every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imetelstat sodium

INTERVENTIONS:
Drug: imetelstat sodium — Given IV
  Other Names: GRN163L; telomerase inhibitor GRN163L

SUMMARY:
This molecular biology and phase II trial studies how well imetelstat sodium works in treating younger patients with recurrent or refractory brain tumors. Imetelstat sodium may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* Molecular Biology:

I. To test the ability of imetelstat (GRN163L) to inhibit telomerase activity by Telomere Repeat Amplification Protocol (TRAP) in tumor and peripheral blood mononuclear cells (PBMNCs) of children with recurrent or refractory HGG or ependymoma.

II. To characterize the pharmacokinetics of imetelstat in plasma, cerebrospinal fluid (CSF), and tumor tissue of children with recurrent or refractory HGG or ependymoma.

* Phase II:

I. To estimate the sustained objective response rates (complete response (CR) plus partial response (PR), sustained for at least 6 weeks) to imetelstat administered intravenously on Days 1 and 8 of a 21-day course at the recommended Phase II pediatric dose, 285mg/m2, in children with recurrent or refractory HGG, ependymoma or DIPG. Independent estimates of the objective response rates will be made for each of the three strata, two of which are histologically defined.

SECONDARY OBJECTIVES:

* Phase II only:

I. To assess evidence of telomerase expression by detection of hTERT mRNA and TERC RNA levels by quantitative reverse transcription polymerase chain reaction (qRT-PCR) and telomerase activity by TRAP in archival tumor tissue (for HGG, and ependymoma strata) and to explore association of telomerase positivity with objective response and progression-free survival (PFS).

II. To estimate the stratum-specific PFS distributions of children with recurrent or refractory HGG, ependymoma or DIPG treated with imetelstat.

* Molecular Biology and Phase II:

I. To characterize the plasma and CSF pharmacokinetics of imetelstat in children with recurrent or refractory HGG, ependymoma or DIPG.

II. To assess evidence of telomerase expression by detection of hTERT mRNA and TERC RNA levels by qRT-PCR, telomerase activity by TRAP, and telomere length by telomere terminal restriction fragment (TRF) analysis in PBMNCs prior to treatment with imetelstat and to assess evidence of telomerase inhibition by TRAP and telomere shortening by TRF analysis serially on treatment with imetelstat.

III. To compare incidence of Alternative Lengthening of Telomeres (ALT) mechanism in pediatric HGG, or ependymoma as determined by four different assays 1) ATRX/DAXX nuclear localization by immunofluorescence (IF) assay; 2) telomere-specific signal by fluorescence in situ hybridization (FISH); 3) telomeric terminal restriction fragment (TRF) analysis by Southern blot; and 4) by C circle assay and to assess correlation of these methods for ALT detection.

IV. To assess whether ALT status is associated with objective response rates for children with recurrent or refractory HGG, or ependymoma treated with imetelstat.

V. To describe MRI characteristics and diffusion changes of recurrent or refractory HGG, ependymoma and DIPG tumors prior to and after treatment with imetelstat to assess for an early diffusion indicator of response.

VI. To measure telomere length of tumors in children with recurrent or refractory HGG, or ependymoma and to assess association of tumor length with tumor response to imetelstat treatment.

VII. To assess hTERT promoter mutations and methylation, H3F3A, ATRX, and DAXX mutations, and examine the effects of these modifications in children with recurrent brain tumors using targeted gene, exome, RNA sequencing and methylation arrays of targeted genomic regions.

OUTLINE:

Molecular Biology Phase: Patients will receive one infusion of imetelstat prior to surgery. Surgery will take place 12-24 hours after the infusion of imetelstat. Patients will continue to receive therapy on the same schedule as the Phase II patients starting 14-21 days after surgery.

Phase II: Patients receive imetelstat sodium IV over 2 hours on days 1 and 8. Treatment repeats every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
INCLUSION CRITERIA:

* MOLECULAR BIOLOGY STUDY

  * Tumor: Histologically confirmed Dx of ependymoma or HGG (such as anaplastic astrocytoma, glioblastoma, gliosarcoma, or anaplastic oligodendroglioma) that is recurrent or refractory to conventional therapy.
  * Subjects must have clinical indications for surgical resection and be amenable to receiving imetelstat prior to tumor resection. Subjects who require emergent surgery are not eligible for the Molecular Biology study.
  * Subjects must provide, fresh flash frozen tumor samples (target 50 mg tissue; as low as 20 mg is adequate) from the time of diagnosis or previous recurrence for the assessment of tumor telomerase activity by the TRAP assay.
* PHASE II STUDY

  * Tumor: Subjects must have recurrent or refractory disease with a histological Dx from either the initial presentation or at the time of recurrence. The requirement for histologic verification is waived for subjects with DIPG (stratum D). The following diagnoses are eligible and will be treated in separate strata (B-D): (B) recurrent or refractory high-grade glioma, (such as anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, anaplastic oligodendroglioma); (C) recurrent or refractory ependymoma; (D) recurrent or refractory DIPG (diagnosis by imaging characteristics acceptable; no histologic confirmation required)
  * Slides from either initial Dx or relapse must be available for central pathology review for Strata B-C. Tissue slides must be sent per Section 10.1. If tissue slides are unavailable, the study chair must be notified prior to study enrollment.
  * All subjects must have bi-dimensionally measurable disease in the brain and/or spine, defined as at least one lesion that can be accurately measured in at least two planes in order to be eligible for this study. Subjects who are enrolled on the Molecular Biology trial and who have measurable disease after the surgical resection and meet all other eligibility criteria for the Phase II study will be counted towards the accrual of the Phase II study.
* FOR BOTH MOLECULAR BIOLOGY AND PHASE II STUDIES

  * Subjects with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration; a baseline detailed neurological exam should clearly document the neurological status of the subject at the time of registration on the study
  * Karnofsky >= 50% for > 16 years of age; Lansky >= 50% for children < 16 years of age documented within 14 days of study registration and within 7 days of the start of study drug administration
  * Hemoglobin >= 8 g/dL (may receive blood transfusions)
  * Absolute neutrophil count > 1,000/ul
  * Platelet count >= 100,000/ul (transfusion independent defined as no platelet transfusions with a 4 week period prior to enrollment)
  * Serum bilirubin < 2.0 mg/dL (patients with Gilbert syndrome, serum bilirubin < 3.0 x upper limit of normal [ULN])
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x institutional ULN
  * Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
  * Alkaline phosphatase < 2.5 x institutional ULN
  * Albumin >= 2 g/dL
  * Adequate coagulation defined as activated partial thromboplastin time (aPTT) < 1.2 x ULN
  * Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:
* Age 1 to < 2 years: maximum serum creatinine (mg/mL) 0.6 for males and 0.6 for females
* Age 2 to < 6 years: maximum serum creatinine (mg/mL) 0.8 for males and 0.8 for females
* Age 6 to < 10 years: maximum serum creatinine (mg/mL) 1 for males and 1 for females
* Age 10 to < 13 years: maximum serum creatinine (mg/mL) 1.2 for males and 1.2 for females
* Age 13 to < 16 years: maximum serum creatinine (mg/mL) 1.5 for males and 1.4 for females
* Age >= 16 years: maximum serum creatinine (mg/mL) 1.7 for males and 1.4 for females
* The threshold creatinine values were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the Centers for Disease and Control (CDC)

  * Subjects on systemic anticoagulants are excluded from this study as the drug can cause minor, transient changes in aPTT
  * Female subjects of childbearing potential must not be pregnant or breast-feeding; female subjects of childbearing potential must have a negative serum or urine pregnancy test; (pregnancy test must be repeated within 48 hours prior to the start of therapy)
  * Subjects of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study
  * Subjects must have recovered from the acute toxicities of all prior therapy before entering this study; for those acute baseline adverse events attributable to prior therapy, recovery is defined as a toxicity grade =< 2, using Common Terminology Criteria for Adverse Events (CTCAE) v.4.0, unless otherwise specified in the Inclusion and Exclusion Criteria
  * Subjects must have received their last dose of known myelosuppressive anticancer chemotherapy at least three (3) weeks prior to study registration or at least six (6) weeks if nitrosourea
  * Subjects must have received their last dose of investigational or biologic agent >= 7 days prior to study registration; in the event that a subject has received an investigational or biologic agent and has experienced >= grade 2 myelosuppression, then at least three (3) weeks must have elapsed prior to registration; if the investigational or biologic agent has a prolonged half-life (>= 7 days) then at least three (3) weeks must have elapsed prior to registration
  * Subjects must have completed at least 3 half-life periods from the last dose of monoclonal antibody prior to registration; Note: A list of half-lives of commonly used monoclonal antibodies is available on the Pediatric Brain Tumor Consortium (PBTC) website under Generic Forms and Templates
  * Subjects must have received their last dose of radiation (XRT):
* 2 weeks prior to study registration for local palliative XRT (small volume)
* 3 months prior to study registration for craniospinal XRT
* 6 weeks (wks) prior to study registration for other substantial bone marrow irradiation

  * Subject must be >= 3 months since autologous bone marrow/stem cell transplantation prior to registration
  * Subjects who are receiving a corticosteroid, such as dexamethasone, must be on a stable or decreasing dosage for at least 1 week prior to registration
  * At least 7 days since the completion of therapy with a hematopoietic growth agent (filgrastim, sargramostim, and erythropoietin) and 14 days for long-acting formulations
  * Ability to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Subjects must not be receiving any other investigational agents
* Subjects with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to imetelstat
* Known coagulopathy or bleeding diathesis
* Subjects with imaging evidence of CNS hemorrhage on baseline MRI obtained within 14 days prior to study enrollment are not eligible; Note: The presence of small punctate areas consistent with hemorrhage will not exclude subjects from participation
* Use of systemic anticoagulant medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, cirrhosis or psychiatric illness/social situations that would limit compliance with study requirements

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (11):
- United States (11):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital- Chicago, Chicago, Illinois
  - NCI - Pediatric Oncology Branch, Bethesda, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Other PBTC investigators can develop a concept proposal and submit it to the PBTC Scientific Committee for a decision to share data and to what extent to share it.

RESULTS

PARTICIPANT FLOW:
Groups:
- Molecular Biology Stratum-A: This is the Molecular Biology arm for Medulloblastoma/PNET Patients
- Molecular Biology Stratum-B: This is the Molecular Biology arm for High-Grade Glioma Patients
- Molecular Biology Stratum-C: This is the Molecular Biology arm for Ependymoma Patients
- Stratum-A: This is the Phase-II stratum for Recurrent or Refractory Medulloblastoma/PNET Patients
- Stratum-B: This is the Phase-II stratum for Recurrent or refractory high-grade glioma patients
- Stratum-C: This is the Phase-II stratum for Recurrent or refractory ependymoma patients
- Stratum-D: This is the Phase-II stratum for Recurrent or refractory diffuse intrinsic pontine gliomas (DIPG) patients
Period: Overall Study
Arm/Group | Molecular Biology Stratum-A | Molecular Biology Stratum-B | Molecular Biology Stratum-C | Stratum-A | Stratum-B | Stratum-C | Stratum-D
Started | 1 | 1 | 1 | 9 | 18 | 4 | 9
Completed | 1 | 1 | 0 | 8 | 18 | 4 | 8
Not Completed | 0 | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Did not receive study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Patient declared ineligible | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Patient inevaluable to start therapy | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Molecular Biology Stratum-A | Molecular Biology Stratum-B | Stratum-A | Stratum-B | Stratum-C | Stratum-D | Total
Number analyzed (Participants) | 1 | 1 | 8 | 18 | 4 | 8 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.41 (NA) — Only one patient | 11.33 (NA) — Only one Patient | 7.94 (4.31) | 11.66 (5.24) | 11.51 (3.84) | 10.45 (2.14) | 10.62 (4.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 7 | 2 | 4 | 15
  Male | 1 | 1 | 6 | 11 | 2 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Numver of Patients With Telomerase-positive Archival Tumors Who Demonstrate at Least 50% Reduction
Description: This outcome measure is for the Molecular biology study only. The assessment was done to identify cases with at least 50% reduction in telomerase activity.
Time Frame: Up to 30 days
Population: This outcome measure is only for the molecular biology study. Telomerase inhibition was assessed and the inhibition level was compared with the baseline level to identify increased inhibition.
Measure: Count of Participants; unit: Participants
Groups:
- Molecular Biology Study: Molecular Biology Phase: Patients will receive one infusion of imetelstat prior to surgery. Surgery will take place 12-24 hours after the infusion of imetelstat. Patients will continue to receive therapy on the same schedule as the Phase II patients starting 14-21 days after surgery.
  Phase II: Patients receive imetelstat sodium IV over 2 hours on days 1 and 8. Treatment repeats every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  imetelstat sodium: Given IV
Arm/Group | Molecular Biology Study
Number analyzed (Participants) | 2
Participants | 1

2. Primary Outcome: Phase II: Stratum-specific Objective Response (CR+PR) Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=50% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR sustained for at least 6 weeks.
  For each stratum separately exact confidence interval estimates will be provided for the true, unknown rates of objective response. Estimated by cumulative incidence functions.
Time Frame: 6 months
Population: This is the Phase-II study cohort, excluding the molecular study patients.
Measure: Count of Participants; unit: Participants
Groups:
- Stratum-D: This is the Phase-II stratum for Recurrent or refractory diffuse intrinsic pontine glioma patients
Arm/Group | Stratum-A | Stratum-B | Stratum-C | Stratum-D
Number analyzed (Participants) | 8 | 18 | 4 | 8
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Telomerase Inhibition
Description: This outcome measure is applicable only for the Molecular biology study arm. Telomerase inhibition was assessed in PBMCs and summarised as 'yes-inhibited' vs. 'no inhibition'
Time Frame: Up to 30 days
Population: Samples from six patients were consequently considered evaluable and were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Molecular Biology Study
Number analyzed (Participants) | 6
Participants | 5

4. Secondary Outcome: Stratum-specific Progression-free Survival (PFS) (Phase II)
Description: Kaplan-Meier estimates of distributions of survival and PFS for all eligible subjects who received at least one dose of imetelstat will be provided separately.
Time Frame: Up to 2 years, from the date of initial treatment to the earliest date of disease progression, second malignancy or death for subjects who fail; and to the date of last contact for subjects who remain at risk for failure, assessed up to 3 years
Population: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Measure: Mean (Standard Error); unit: days
Arm/Group | Stratum-A | Stratum-B | Stratum-C | Stratum-D
Number analyzed (Participants) | 8 | 18 | 4 | 8
days | 30 (3.06) | 54.2 (9.97) | 50.3 (16.25) | 52.6 (14.50)

5. Secondary Outcome: Number of Patients With Telomerase Expression Data by Detection of hTERT mRNA and TERC RNA Levels by qRT-PCR and Telomerase Activity by TRAP in Archival Tumor Tissue and to Explore Association of Telomerase Positivity With Objective Response and PFS
Description: This secondary objective is for Stratum-B and C only, which enroll HGG and ependymoma patients. We will describe the evidence of telomerase expression by detection of hTERT mRNA and TERC RNA levels by qRT-PCR and telomerase activity by TRAP in archival tumor tissue; Association of telomerase positivity with objective response and PFS will not be able to be conducted as the study was terminated early and there was no objective response.
Time Frame: Up to 30 days. Due to small number of patients evaluable for this objective, we can only provide number of patients with the targetted markers as no analysis with PFS is possible.
Population: This objective is for STRATUM-C patients only, having only 4 patients with TRAP, TERT and TERC levels measured. Due to small sample and having no objective response, association studies of these markers with Objective Reponse and PFS were not possible. Therefore, we only report the the percentage of cases with at least weak TRAP activity.
Measure: Count of Participants; unit: Participants
Groups:
- Stratum-C: This objective is for HGG and ependymoma patients only.
Arm/Group | Stratum-C
Number analyzed (Participants) | 4
Participants
  TRAP | 3
  TERT | 3
  TERC | 3

6. Secondary Outcome: Quantitative MRI Parameters of Tumors Prior to and After Treatment With Imetelstat (Molecular Biology and Phase II Studies)
Description: This outcome measure was for both Molecular biology and Phase II studies. We will not be able to present the results of this objective as the study was terminated early.
Time Frame: Up to 30 days
Population: This study has been terminated early and the study team decided not to pursue this aim as the results would be inconclusive due to small sample size. Neither the neuroimaging, nor the biology data are available for these patients.
Groups:
- Treatment (Imetelstat Sodium): Molecular Biology Phase: Patients will receive one infusion of imetelstat prior to surgery. Surgery will take place 12-24 hours after the infusion of imetelstat. Patients will continue to receive therapy on the same schedule as the Phase II patients starting 14-21 days after surgery.
  Phase II: Patients receive imetelstat sodium IV over 2 hours on days 1 and 8. Treatment repeats every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  imetelstat sodium: Given IV
Arm/Group | Treatment (Imetelstat Sodium)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years, which is the total possible therapy duration.
Description: The AEs we report were experienced while the participants were on study.
Groups:
- Molecular Study-A: Molecular Study arm for Recurrent or Refractory Medulloblastoma/PNET Patients
- Molecular Study-B: Molecular Study arm for Recurrent or refractory high-grade glioma patients
Arm/Group | Molecular Study-A | Molecular Study-B | Stratum-A | Stratum-B | Stratum-C | Stratum-D
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 3/8 | 4/18 | 2/4 | 3/8
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 8/8 | 16/18 | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molecular Study-A (N=1) | Molecular Study-B (N=1) | Stratum-A (N=8) | Stratum-B (N=18) | Stratum-C (N=4) | Stratum-D (N=8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify[Death due to pr (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify[Progressive dis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify[Cervical hemorrhage] (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify[increased secretions requiring freq (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death, NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molecular Study-A (N=1) | Molecular Study-B (N=1) | Stratum-A (N=8) | Stratum-B (N=18) | Stratum-C (N=4) | Stratum-D (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (4) | 7 (7) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify[Diplopia] (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scleral disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 4 (4) | 4 (4) | 1 (1) | 3 (3)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 4 (4) | 8 (8) | 0 (0) | 6 (6)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 4 (4) | 7 (7) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify[increased PT] (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 5 (5) | 8 (8) | 0 (0) | 6 (6)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 4 (4) | 9 (9) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 8 (8) | 11 (11) | 1 (1) | 5 (5)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 8 (8) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify[Foot pain] (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 2 (2)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify[Inability to tolerate own secretions] (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify[Urinary Hesitancy] (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No